CLINICAL TRIAL: NCT01313169
Title: Electronic Medical Record Reminders and Panel Management to Improve Primary Care of Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Donald W. Reynolds Foundation (Other)
Responsible Party: Principal Investigator, Timothy S. Loo, Assistant Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2009P000108
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: EMR Reminders to Improve Rates of Recommended Care
Keywords: Electronic medical record reminders, Panel management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- EMR reminder (Experimental): EMR reminder
  Interventions: Other: EMR Reminder
- EMR reminder + Panel management (Experimental): EMR reminder + Panel manager
  Interventions: Other: EMR Reminder + Panel management
- Control (No Intervention): Control

INTERVENTIONS:
Other: EMR Reminder — EMR reminders displayed
  Arms: EMR reminder
Other: EMR Reminder + Panel management — EMR Reminder + Panel management
  Arms: EMR reminder + Panel management

SUMMARY:
The investigators conducted a controlled trial to assess the effectiveness of electronic medical record (EMR) reminders, with or without a panel manager, on completion of health care proxy, osteoporosis screening, and influenza and pneumococcal vaccinations for patients age 65 or older. The investigators hypothesized that EMR reminders would improve adherence to practice guidelines and that benefits would be enhanced with the support of a panel manager.

ELIGIBILITY:
Inclusion Criteria:

* All practicing faculty primary care physicians at Beth Israel Deaconess Medical Center General Medicine & primary care ambulatory clinic

Exclusion Criteria:

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2009-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
a designated health care proxy | 12 months after intervention made available
  A designated health care proxy was defined as a verified proxy documented in the EMR's health care proxy field
initial bone density scan | 12 months after intervention made available
  The initial bone density scan measure was defined as having either bone density scan ordered or a bone density scan completed
administration of annual influenza vaccine | 12 months after intervention started
  Administration of influenza vaccine was defined as vaccine documented as given at any location
administration of pneumococcal vaccine | 12 months after the start of the intervention
  Administration of pneumococcal vaccine was defined as vaccine documented as given at any location.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Loo, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Loo TS, Davis RB, Lipsitz LA, Irish J, Bates CK, Agarwal K, Markson L, Hamel MB. Electronic medical record reminders and panel management to improve primary care of elderly patients. Arch Intern Med. 2011 Sep 26;171(17):1552-8. doi: 10.1001/archinternmed.2011.394. PMID 21949163